CLINICAL TRIAL: NCT03118362
Title: Clearance of Acetate During Fluid Resuscitation of Critically Ill Burn Patients: The CARE Trial.
Brief Title: Fluid Resuscitation in Burn Patients
Acronym: CARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P160502
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Severe Burns; Fluid Resuscitation
Keywords: Burns; Critically ill; Acid-Base status
MeSH Terms: conditions — Burns; Critical Illness | interventions — Plasmalyte A; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Plasmalyte® is a balanced solution containing a low chloride concentration (i.e. 98 mmol/L) which may overcome overwhelm the potential risks associated with hyperchloremic solutions. Plasmalyte® also contains acetate (27 mmol/L) and gluconate (23 mmol/L) as buffer solutions.
  Ringer Lactate® is also a balanced solution containing a low chloride concentration (i.e. 111 mmol/L)
Who Masked: Participant
Masking Description: the crystalloid infusion solutions will be introduce in Opabag
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasmalyte® (Experimental): Plasmalyte® is a balanced solution containing a low chloride concentration (i.e. 98 mmol/L), it also contains acetate (27 mmol/L) and gluconate (23 mmol/L) as buffer solutions.
  Interventions: Drug: Plasmalyte
- Ringer Lactate® (Experimental): Ringer Lactate® is a balanced solution containing a low chloride concentration (i.e. 111mmol/L), it also contains lactate (29 mmol/L) as buffer solutions.
  Interventions: Drug: Ringer lactate

INTERVENTIONS:
Drug: Plasmalyte — Parenteral administration of Plasmalyte initiated immediately after inclusion at a dosage of 4 ml / kg per percentage area of skin burned for the first 24 hours after burn injury and adjusted based on hemodynamic monitoring.
  Each patient will receive this solution up to 5 days.
  Other Names: PLASMALYTE VIAFLO
  Arms: Plasmalyte®
Drug: Ringer lactate — Parenteral administration of Ringer lactate initiated immediately after inclusion at a dosage of 4 ml / kg per percentage area of skin burned for the first 24 hours after burn injury and adjusted based on hemodynamic monitoring.
  Each patient will receive this solution up to 5 days.
  Other Names: RINGER LACTATE VIAFLO
  Arms: Ringer Lactate®

SUMMARY:
Balanced solutions with low chloride concentration could represent an alternative to high chloride concentration solutions. Such balanced solutions contain other acid as buffers (i.e. acetate and/or gluconate). However, acetate has been associated with alteration of cardiac function when used as buffer in dialysate when high acetate concentrations are used and could promote the development of metabolic acidosis if it accumulates. Therefore, the safety of such solutions remains poorly explored. Because critically ill patients receive large amount of fluid during the early phase of resuscitation, large amount of acetate are to be administrated if such solutions are used. While acetate-containing solutions have been suggested to be safe in this setting, studies are still lacking regarding clearance and accumulation in critically ill patients.

It is expected to include 28 patients, the objective to analyze the data of 20 patients.

DETAILED DESCRIPTION:
The main objectives of the study is 1) to determine whether Plasmalyte® promote the development of metabolic acidosis in comparison with an acetate-free balanced solutions: Ringer lactate (chloride concentration of 111 mmol/L) and 2) to determine Acetate & gluconate clearance during fluid resuscitation of severely burn patients Plasmalyte® (chloride concentration of 98 mmol/L) . Severely burn patients will be randomized to receive Plasmalyte® or Ringer Lactate for initial fluid resuscitation during the first 5 days following admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* TBSA>30%
* Admission to an intensive care unit within 12 hours after burn injury
* Signed informed consent to Patient / Parent / ( Inclusion in Emergency and Consent is Collected)
* social Insurance cover

Exclusion Criteria:

* Decline to participate
* pregnancy
* Metabolic alkalosis (excess of base> 5mmol / L)
* legal obstacle to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
The main endpoint is to compare the base deficit in patients receiving Plasmalyte® or Ringer lactate after 24 hours of admission. | after 24 hours of admission.
  Arterial blood gas analysis

SECONDARY OUTCOMES:
Acetate, gluconate and lactate clearance respectively in patients receiving Plasmalyte® or Ringer lactate. | Every 6 hours for 48 hours, then every 12 hours for acid-base status during 5 days.
  Arterial blood gas analysis
acid-base status and strong ion difference after 24 hours of Plasmalyte® or Ringer lactate infusion | Every 6 hours for 48 hours, then every 12 hours for acid-base status during 5 days.
  Arterial blood gas analysis
Occurrence of cardiac dysfunction, defined as altered left ventricular ejection fraction(<50%) | Every day during 5 days
  Trans-thoracic or trans-esophageal ultrasound
Incidence of AKI (according to the KDIGO definition) | Every day during 5 days
  urine output and serum creatinine
Sequential Organ Failure Assessment score | During the first 5 days of intensive care unit stay
  SOFA score calculation
mortality at day 28 | At 28 day after admission
  Mortality will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Legrand, MD, PhD, Principal Investigator — Departement of Anesthesiology, Critical Care and Burn Unit; Saint-Louis hospital, 1 Avenue Claude Vellefaux, 75010, Paris & University Paris Diderot
Locations (1):
- Departement of Anesthesiology, Critical Care and Burn Unit; Saint-Louis hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn RG. Should anaesthetists stop infusing isotonic saline? Br J Anaesth. 2014 Jan;112(1):4-6. doi: 10.1093/bja/aet292. No abstract available. PMID 24318694
- [Background] Shaw AD, Bagshaw SM, Goldstein SL, Scherer LA, Duan M, Schermer CR, Kellum JA. Major complications, mortality, and resource utilization after open abdominal surgery: 0.9% saline compared to Plasma-Lyte. Ann Surg. 2012 May;255(5):821-9. doi: 10.1097/SLA.0b013e31825074f5. PMID 22470070
- [Background] Zhou F, Peng ZY, Bishop JV, Cove ME, Singbartl K, Kellum JA. Effects of fluid resuscitation with 0.9% saline versus a balanced electrolyte solution on acute kidney injury in a rat model of sepsis*. Crit Care Med. 2014 Apr;42(4):e270-8. doi: 10.1097/CCM.0000000000000145. PMID 24335444
- [Background] Davies PG, Venkatesh B, Morgan TJ, Presneill JJ, Kruger PS, Thomas BJ, Roberts MS, Mundy J. Plasma acetate, gluconate and interleukin-6 profiles during and after cardiopulmonary bypass: a comparison of Plasma-Lyte 148 with a bicarbonate-balanced solution. Crit Care. 2011;15(1):R21. doi: 10.1186/cc9966. Epub 2011 Jan 14. PMID 21235742
- [Background] Morgan TJ, Power G, Venkatesh B, Jones MA. Acid-base effects of a bicarbonate-balanced priming fluid during cardiopulmonary bypass: comparison with Plasma-Lyte 148. A randomised single-blinded study. Anaesth Intensive Care. 2008 Nov;36(6):822-9. doi: 10.1177/0310057X0803600611. PMID 19115651